CLINICAL TRIAL: NCT03259529
Title: A Phase I/II Clinical Trial to Evaluate the Safety and Efficacy of Bendamustine, Gemcitabine, Rituximab, Nivolumab Combination (BeGeRN) in Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma
Brief Title: Safety and Efficacy of Bendamustine, Gemcitabine, Rituximab, Nivolumab (BeGeRN) in Patients With r/r DLBCL
Acronym: BeGeRN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Vice-director for science of R.M. Gorbacheva Memorial Institute of Hematology, Oncology and Transplantation, St. Petersburg State Pavlov Medical University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DLBCL BeGeRN 1/2
Record Dates: First submitted 2017-08-22; First posted 2017-08-23 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Diffuse Large B-cell Lymphoma; Nivolumab; Bendamustine Hydrochloride; Gemcitabine; Rituximab
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Bendamustine Hydrochloride; Gemcitabine; Nivolumab; Rituximab

STUDY DESIGN:
Intervention Model Description: There will be 2 parts in this study. In Part 1, the safety of combination treatment will be evaluated prior to expansion of enrollment to evaluate treatment effect in Part 2. The arms in Part 1 include 3 different dosage regimens of gemcitabine (500 / 700 / 1000). Part 2 of the study will further characterize the safety and evaluate the antitumor activity of drug combination by enrolling patients at the recommended dose schedule determined in Part 1.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gemcitabine 500 (Experimental): Days 1,2 Bendamustine Hydrochloride 70 mg/m2/day iv; Days 1,8,15 Gemcitabine 500 mg/m2/day iv; Days 1,15 Nivolumab 1mg/kg/day iv; Day 0 Rituximab 375mg/kg/day iv.
  Duration of cycle 28 days
  Interventions: Drug: Bendamustine hydrochloride; Drug: Gemcitabine 500 mg; Drug: Nivolumab; Drug: Rituximab
- Gemcitabine 700 (Experimental): Days 1,2 Bendamustine Hydrochloride 70 mg/m2/day iv; Days 1,8,15 Gemcitabine 700 mg/m2/day iv; Days 1,15 Nivolumab 1mg/kg/day iv; Day 0 Rituximab 375mg/kg/day iv.
  Duration of cycle 28 days
  Interventions: Drug: Bendamustine hydrochloride; Drug: Gemcitabine 700 mg; Drug: Nivolumab; Drug: Rituximab
- Gemcitabine 1000 (Experimental): Days 1,2 Bendamustine Hydrochloride 70 mg/m2/day iv; Days 1,8,15 Gemcitabine 1000 mg/m2/day iv; Days 1,15 Nivolumab 1mg/kg/day iv; Day 0 Rituximab 375mg/kg/day iv.
  Duration of cycle 28 days
  Interventions: Drug: Bendamustine hydrochloride; Drug: Gemcitabine 1000 mg; Drug: Nivolumab; Drug: Rituximab

INTERVENTIONS:
Drug: Bendamustine hydrochloride — 70 mg/m2 by intravenous (IV) infusion for up to 2 cycles
  Other Names: Ribomustin
Drug: Gemcitabine 500 mg — 500 mg/m2 by intravenous (IV) infusion on day 1,8,15 for up to 2 cycles
  Other Names: Gemzar
  Arms: Gemcitabine 500
Drug: Gemcitabine 700 mg — 700 mg/m2 by intravenous (IV) infusion on day 1,8,15 for up to 2 cycles
  Other Names: Gemzar
  Arms: Gemcitabine 700
Drug: Gemcitabine 1000 mg — 1000 mg/m2 by intravenous (IV) infusion on day 1,8,15 for up to 2 cycles
  Other Names: Gemzar
  Arms: Gemcitabine 1000
Drug: Nivolumab — 1 mg/kg by intravenous (IV) infusion on day 1,15 for up to 2 cycles
  Other Names: Opdivo
Drug: Rituximab — 375 mg/m2 by intravenous (IV) infusion on day 0 for up to 2 cycles

SUMMARY:
Despite the current advances in clinical oncology, the prognosis of patients with resistant diffuse large B cell lymphoma or relapse after high dose chemotherapy is dismal. Therefore there is a need for the introduction of novel treatment regimens. This phase I/II trial evaluates the safety and efficacy of combination bendamustine, gemcitabine, nivolumab and rituximab in patients with relapsed or refractory diffuse large B-cell lymphoma. The safety of combination treatment will be evaluated with the determination of recommended dose schedule prior to expansion of enrollment to evaluate the antitumor activity of bendamustine, gemcitabine, rituximab, and nivolumab.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Histologically confirmed diffuse large B-cell lymphoma
* Refractory or relapsed after at least two prior lines of treatment (i.e. induction and salvage regimen) for diffuse large B-cell lymphoma.
* Age 18-70 years old
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2
* Signed informed consent
* No severe concurrent illness

Exclusion Criteria:

* Uncontrolled bacterial or fungal infection at the time of enrollment
* Requirement for vasopressor support at the time of enrollment
* Karnofsky index <30%
* Pregnancy
* Somatic or psychiatric disorder making the patient unable to sign informed consent
* Active or prior documented autoimmune disease requiring systemic treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
The recommended phase 2 dose (RP2D) | 6 months
  The recommended phase 2 dose (RP2D) of Bendamustine Hydrochloride and Gemcitabine in combination with Nivolumab and Rituximab in patients with Diffuse Large B-cell Lymphoma
Overall Response Rate (ORR) | 12 months
  Overall response rate (ORR), defined as the proportion of patients with complete response (CR) or partial response (PR) in measurable lesions as defined by LYRIC criteria and duration of response.

SECONDARY OUTCOMES:
Frequency of grade 3 or higher treatment-related adverse events by CTCAE 4.03 | 12 months
  Toxicity parameters based on NCI CTCAE 4.03 grades: hematological toxicity (CBC), hepatotoxicity (liver function tests), nephrotoxicity (creatinine), neurotoxicity (attending physician assessment), fatigue (attending physician assessment), rash (attending physician assessment), colitis (attending physician assessment), pneumonitis (attending physician assessment), autoimmune disorders (level of hormones, presence of autoimmune antibodies, attending physician assessment).
Duration of Response (DOR) | 12 months
Progression-Free Survival (PFS) | 12 months
Overall Survival (OS) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Boris V Afanasyev, Ph.D, Principal Investigator — St. Petersburg State Pavlov Medical University
Locations (1):
- First Pavlov State Medical University of St. Petersburg, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided